CLINICAL TRIAL: NCT00262353
Title: Elimination of Protein-bound Uremic Retention Solutes by Prometheus Artificial Hepatic System Versus Conventional Dialysis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study never started because of safety alerts in literature regarding the topic to be examined
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2004/416
Record Dates: First submitted 2005-12-04; First posted 2005-12-06 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-07

CONDITIONS: Renal Failure, Chronic
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Dialysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Dialysis with different artificial devices

SUMMARY:
Comparison of the efficacy of dialysis by conventional dialysis versus Prometheus artificial hepatic system

DETAILED DESCRIPTION:
After inclusion, patients will be dialysed with low-flux artificial kidneys. 1 week of dialysis exists of 3 days of dialysis. In week 4, day 2, patients will be treated once with the Prometheus artificial hepatic system or with high-flux dialysis. The other days low-flux kidneys will be used. Week 5 and 6 are a wash-out period. Week 7 is identical to week 4 but the other system than in week 4 is used. Blood samples are taken at regular moments in week 3, week 4 (day 2) and week 7 (day 2).

ELIGIBILITY:
Inclusion Criteria:

* Stable patients
* At least 3 months on dialysis
* Arterio-venous fistula

Exclusion Criteria:

* Diabetic patients
* Malignancies
* Acute illnesses

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Determination of the concentration of protein-bound toxins after treatment with different artificial devices

SECONDARY OUTCOMES:
Determination of the kinetics of protein-bound toxins after treatment with different artificial devices

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Vanholder, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website of the University Hospital Ghent — http://www.uzgent.be